CLINICAL TRIAL: NCT03919669
Title: Longitudinal Evaluation of [18-F]MK-6240 as a Novel Tau PET Radiotracer in Patients With Alzheimer's Disease Dementia or Mild Cognitive Impairment Compared to Healthy Volunteers
Brief Title: A Longitudinal Evaluation of a Radiotracer for Use in Tau Tracking
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Cerveau Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018-1348; A534255 (Other: UW Madison); SMPH/MEDICINE/GER-AD DEV (Other: UW Madison); Protocol Version 8/26/2021 (Other: UW Madison)
Record Dates: First submitted 2019-04-15; First posted 2019-04-18 (Actual); Results first posted 2023-08-03 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- All Subjects (Experimental): All subjects will complete PET imaging sessions evaluating the tau PET radioligand [18F]MK-6240 at baseline, as well as at 6, 12 and 24 months post-baseline.
  If unable to complete the 6 month, 12 month, or 24 month visit, an 18 month and/or 30 month visit may instead be scheduled, totaling a maximum of four time points.
  Interventions: Drug: All Subjects

INTERVENTIONS:
Drug: All Subjects — All subjects will be given the experimental tau PET radioligand [18F]MK-6240

SUMMARY:
This is a longitudinal, observational study evaluating the imaging characteristics of the tau PET radioligand [18F]MK-6240 in Alzheimer's disease (AD), Mild Cognitive Impairment (MCI) and Healthy Volunteer (HV) subjects. Up to 42 subjects, including approximately 28 MCI/mild AD subjects, up to 5 moderate AD subjects, and 9 similarly aged HV subjects will be consented and screened. Imaging procedures include [11C]PiB to evaluate amyloid deposition, [18F]MK-6240 PET, and structural MRI. All subjects complete an evaluable baseline [18F]MK-6240 PET scan, as well as scans at 6, 12 and 24 months post-baseline. If unable to complete the 6 month, 12 month, or 24 month visit, an 18 month and/or 30 month visit may instead be scheduled, totaling a maximum of four time points.

ELIGIBILITY:
Inclusion Criteria for all subjects:

* Signed and dated written informed consent must be obtained from the subject to enter the study and before any assessment is performed.
* Pregnancy: Participant is not pregnant at the time of the PET and MRI imaging exams. Urine pregnancy tests will be conducted as needed with pre-menopausal women who are of child-bearing potential.
* Willing and able to undergo study procedures and study schedule
* Availability of a study partner who has frequent and sufficient contact with the subject and is able to provide accurate information regarding the subject's cognitive and functional abilities for the CDR, agrees to accompany the subject and provide information at visits or is available by phone. The study partner must have sufficient cognitive capacity, in the judgment of the investigator, to accurately report upon the subject's behavior and cognitive and functional abilities.
* Healthy with no clinically relevant finding on physical examination at screening and upon reporting for the Baseline [18F]MK-6240 imaging visit.

Inclusion Criteria for Healthy Volunteers

* Normal Cognition based on cognitive results at screening.
* Healthy with no clinically relevant finding on physical examination at screening and upon reporting for the Baseline [18F]MK-6240 imaging visit.
* CDR global score =0

Inclusion Criteria for Subjects with a Diagnosis of MCI or Dementia Due to AD

* Have screening [11C]PiB PET imaging demonstrating amyloid binding based on qualitative read or DVR index value >1.20.
* MMSE score 26-30 (inclusive), CDR global score 0.5 for subjects with MCI
* MMSE score 22-26 (inclusive), CDR global score 0.5 or 1 for subjects with mild dementia due to AD
* MMSE score 16-21 (inclusive), CDR global score 1-2 for subjects with moderate dementia due to AD
* Subjects with MCI must meet 2018 research criteria for MCI (Jack et al., 2018).
* Subjects with dementia must meet 2018 research criteria for dementia (Jack et al., 2018).
* A structural brain MRI with no evidence of non-AD disease to account for dementia or MRI exclusion criteria.

Exclusion Criteria for all subjects

* Lack of capacity to provide informed consent at study entry.
* Subject has received an investigational drug or device within 30 days of screening. Other experimental PET radiotracer drugs are not excluded.
* For women, pregnant, lactating or breastfeeding or intention to become pregnant.
* Evidence of unstable or untreated clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, alternative neurological, immunodeficiency, pulmonary, or other disorder or disease. Stable, treated chronic medical conditions like hypertension, hypercholesterolemia, diabetes mellitus, non-metastatic dermatologic or prostatic cancer, etc. are acceptable as long as they do not, in the study investigator's opinion, contribute to cognitive dysfunction or limit participation in study procedures.
* Any illness or other consideration that makes it unlikely that the subject will be able to complete the 26-month study.
* Current or prior history (within past 5 years) of significant alcohol or substance abuse as determined by the investigator.
* Psychiatric disorders that may interfere with the study including current major Axis I DSM-V disorders including but not limited to severe Major depression, current or history of bipolar I disorder, or schizophrenia.
* Non-English speakers or subjects who are unable to comprehend study materials are excluded at entry
* MRI exclusion criteria include: Findings that may be responsible for neurologic status of the subject such as significant evidence of cerebrovascular disease with multiple infarcts, infectious disease, space-occupying lesion, normal pressure hydrocephalus, CNS trauma, or any other structural abnormality that may impact cognition or image analysis, as judged by the investigator.
* MRI-incompatible implants or devices such as certain cardiac pacemakers or defibrillators, insulin pumps, cochlear implants, metallic ocular foreign body, implanted neural stimulators, CNS aneurysm clips and other medical implants that have not been certified for MRI, or history of claustrophobia in MRI that prevents completion of MRI protocol.
* Treatment with any therapeutic molecule that targets Aβ or tau within 12 months prior to screening.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-04-02 (Actual); Primary Completion 2022-05-19 (Actual); Study Completion 2022-05-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Wisconsin-Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Volunteers: As described in the study eligibility criteria:
  * Normal Cognition based on cognitive results at screening.
  * Healthy with no clinically relevant finding on physical examination at screening and upon reporting for the Baseline [18F]MK-6240 imaging visit.
  * CDR global score =0
- Mild Cognitive Impairment: As described in the study eligibility criteria:
  * Have screening [11C]PiB PET imaging demonstrating amyloid binding based on qualitative read or DVR index value >1.20.
  * MMSE score 26-30 (inclusive), CDR global score 0.5 for subjects with MCI
  * MMSE score 22-26 (inclusive), CDR global score 0.5 or 1 for subjects with mild dementia due to AD
  * MMSE score 16-21 (inclusive), CDR global score 1-2 for subjects with moderate dementia due to AD
  * A structural brain MRI with no evidence of non-AD disease to account for dementia or MRI exclusion criteria.
- Dementia: As described in the study eligibility criteria:
  * Have screening [11C]PiB PET imaging demonstrating amyloid binding based on qualitative read or DVR index value >1.20.
  * MMSE score 26-30 (inclusive), CDR global score 0.5 for subjects with MCI
  * MMSE score 22-26 (inclusive), CDR global score 0.5 or 1 for subjects with mild dementia due to AD
  * MMSE score 16-21 (inclusive), CDR global score 1-2 for subjects with moderate dementia due to AD
Period: Overall Study
Arm/Group | Healthy Volunteers | Mild Cognitive Impairment | Dementia
Started | 6 | 8 | 13
Completed | 5 | 8 | 13
Not Completed | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Volunteers | Mild Cognitive Impairment | Dementia | Total
Number analyzed (Participants) | 6 | 8 | 13 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1 | 2
  >=65 years | 5 | 8 | 12 | 25
Age, Continuous [Mean (Full Range); unit: years] | 69.85 [62 to 73] | 71.60 [67 to 78] | 74.52 [59 to 84] | 72.62 [59 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 8 | 13
  Male | 3 | 6 | 5 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 8 | 13 | 27
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 6 | 8 | 13 | 27
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 8 | 13 | 27

OUTCOME MEASURES:

1. Primary Outcome: Change in [18F]MK-6240 Standard Uptake Value Ratio (SUVR) Uptake
Description: Composite mean SUVR across standard regions including: numerator was the entorhinal, amygdala, fusiform, inferior temporal, middle temporal cortex; denominator was the inferior cerebellum cortex. The SUVR is a ratio and has a theoretic interpretable minimum of 1.0. This primary outcome is reported by the three primary groups: Healthy Volunteers, Mild Cognitive Impairment, and Dementia.
Time Frame: Baseline to 12 months
Population: 26 of the 27 participants completed the 12 month interval
Measure: Mean (Standard Deviation); unit: SUVR
Arm/Group | Healthy Volunteers | Mild Cognitive Impairment | Dementia
Number analyzed (Participants) | 6 | 8 | 13
SUVR | 0.00 (0.05) | 0.10 (0.07) | 0.12 (0.16)

2. Secondary Outcome: The Correlation Between the Change in [18F]MK-6240 Uptake and the Change in the Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-cog) Using Items 1-11
Description: This outcome is correlational and therefore the arms/groups are collapsed to All Subjects so that we can assess the overall pattern of relationship between cognition and tau signal across the entire continuum of Alzheimer's disease. The ADAS-cog is one of the most frequently used tests to measure cognition in clinical trials in AD. The first 11 items of the ADAS-cog were used for this outcome. The ADAS was developed as a two-part scale: one that measured cognitive functions and one that measured non-cognitive functions such as mood and behavior. Most current research, including this study, uses the ADAS-Cog, which is the sub-scale that measures cognitive ability. The ADAS-cog score is based on incorrect items or errors and has a range of 0-50, where lower scores indicate better cognitive functioning.
Time Frame: Baseline to 12 months
Population: 26 of the 27 participants completed the 12 month interval
Measure: Number; unit: Spearman Rho
Groups:
- All Subjects: All subjects will complete PET imaging sessions evaluating the tau PET radioligand [18F]MK-6240 at baseline, as well as at 6, 12 and 24 months post-baseline.
  If unable to complete the 6 month, 12 month, or 24 month visit, an 18 month and/or 30 month visit may instead be scheduled, totaling a maximum of four time points.
  All Subjects: All subjects will be given the experimental tau PET radioligand [18F]MK-6240
Arm/Group | All Subjects
Number analyzed (Participants) | 27
Spearman Rho | .02

3. Secondary Outcome: Correlate the Changes in [18F]MK-6240 Uptake and Changes in Clinical Cognitive Assessments by Clinical Dementia Rating Scale (CDR).
Description: This outcome is correlational and therefore the arms/groups are collapsed to All Subjects so that we can assess the overall pattern of relationship between cognition and tau signal across the entire continuum of Alzheimer's disease. The CDR was developed primarily for use in persons with dementia of the Alzheimer type. The six domains of CDR are: Memory, Orientation, Judgment and Problem-solving, Community Affairs, Home and Hobbies, and Personal Care. Each domain is rated on a 5-point scale of functioning: 0 no impairment; 0.5 questionable impairment; 1 mild impairment; 2 moderate impairment; and 3 severe impairment. The Sum of Boxes is the score used which is simply the sum of the 6 Domain Box Scores. The range is 0-18 with lower scores indicating better cognitive function.
Time Frame: Baseline to 12 months
Population: 26 of the 27 participants completed the 12 month interval
Measure: Number; unit: Spearman Rho
Arm/Group | All Subjects
Number analyzed (Participants) | 27
Spearman Rho | .23

4. Secondary Outcome: Correlate the Changes in [18F]MK-6240 Uptake and Changes in Clinical Cognitive Assessments by Mini-Mental Status Exam (MMSE)
Description: This outcome is correlational and therefore the arms/groups are collapsed to All Subjects so that we can assess the overall pattern of relationship between cognition and tau signal across the entire continuum of Alzheimer's disease. The MMSE is a sensitive, valid and reliable 30-point questionnaire that is used extensively in clinical and research settings to measure cognitive impairment. It is commonly used as screening tool for dementia. It is also used to estimate the severity and progression of cognitive impairment and to follow the course of cognitive changes in an individual over time; thus, making it an effective way to document an individual's response to treatment. The range is 0-30 with higher scores indicating better cognitive functioning.
Time Frame: Baseline to 12 months
Population: 26 of the 27 participants completed the 12 month interval
Measure: Number; unit: Spearman Rho
Arm/Group | All Subjects
Number analyzed (Participants) | 27
Spearman Rho | .43

5. Secondary Outcome: Change in [18F]MK-6240 Standard Uptake Value Ratio (SUVR) Uptake
Description: as for outcome 1
Time Frame: Baseline to 24 months
Population: 26 of the 27 participants completed the 24 month interval
Measure: Mean (Standard Deviation); unit: SUVR
Arm/Group | Healthy Volunteers | Mild Cognitive Impairment | Dementia
Number analyzed (Participants) | 6 | 8 | 13
SUVR | -.01 (.09) | .21 (.16) | .24 (.34)

6. Secondary Outcome: Change in [18F]MK-6240 Standard Uptake Value Ratio (SUVR) Uptake
Description: as for outcome 1
Time Frame: Baseline to 6 months
Population: 26 of the 27 participants completed the 6 month interval
Measure: Mean (Standard Deviation); unit: SUVR
Arm/Group | Healthy Volunteers | Mild Cognitive Impairment | Dementia
Number analyzed (Participants) | 6 | 8 | 13
SUVR | -.03 (.04) | -.07 (.26) | .19 (.33)

ADVERSE EVENTS:
Time Frame: Given that this longitudinal study involves procedures that will occur at 6-12 month intervals and does not include chronic treatment with an investigational agent, adverse events (AEs) and serious adverse events (SAEs) were captured during the study visit before and after PiB and MK6240 scans, within 24 hours after the scan. Adverse events were monitored from signing the informed consent form through study completion, on average 2.5 years.
Description: The subjects received a phone call within 4 days from the study team for the purpose of ascertaining their wellbeing and information on adverse events that occur within 24 hours after the scan. If any adverse events were discovered, a clinician continued to follow up with the subject until resolved.
Groups:
- Dementia; Healthy Volunteer; Mild Cognitive Impairment: All subjects will complete PET imaging sessions evaluating the tau PET radioligand [18F]MK-6240 at baseline, as well as at 6, 12 and 24 months post-baseline.
  If unable to complete the 6 month, 12 month, or 24 month visit, an 18 month and/or 30 month visit may instead be scheduled, totaling a maximum of four time points.
  All Subjects: All subjects will be given the experimental tau PET radioligand [18F]MK-6240
Arm/Group | Dementia | Healthy Volunteer | Mild Cognitive Impairment
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/6 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/6 | 0/8
Other Adverse Events (participants affected / at risk) | 3/13 | 1/6 | 0/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dementia (N=13) | Healthy Volunteer (N=6) | Mild Cognitive Impairment (N=8)
Injection Site Reaction (General disorders) | 1 (1) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Infusion Site Extravasation (General disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
This study included a small sample size of 6 healthy volunteers, 8 Mild Cognitive Impairment, and 13 Dementia subjects. This limits the statistical conclusions of the study. The study subjects were all non-hispanic, white participants. This limits the generalizability of the results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-08-26): https://cdn.clinicaltrials.gov/large-docs/69/NCT03919669/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-18): https://cdn.clinicaltrials.gov/large-docs/69/NCT03919669/SAP_001.pdf